CLINICAL TRIAL: NCT01275222
Title: A Phase I-II, Open-label Study of RAD001 in Combination With Glivec®/Gleevec™ (Imatinib) in Patients With Glivec/Gleevec-refractory/Resistant Gastrointestinal Stromal Tumors.
Brief Title: Everolimus in Combination With Imatinib in Patients With Glivec Refractory/Resistant Gastrointestinal Stromal Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001C2206
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Results first posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: RAD001; everolimusGIST; everolimus; mTOR; Imatinib resistant; Imatinib-refractory/resistant; gastrointestinal stromal tumors; Gastrointestinal Stromal Tumors(GIST); soft tissue sarcoma; stomach tumor; tumor of interstitial cells of Cajal (ICC); digestive system cancer
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Sarcoma; Stomach Neoplasms; Digestive System Neoplasms | interventions — Everolimus; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase l: RAD001 20mg/week (Experimental): RAD001 20 mg was given once a week.
  Interventions: Drug: RAD001
- Phase l: RAD001 2.5mg/day + Glivec 600mg/day (Experimental): RAD001 2.5 mg was given in combination with Glivec/Gleevec 600mg/day.
  Interventions: Drug: RAD001; Drug: Imatinib 600mg/day (Glevec is the brand name for imatinib)
- Phase l: RAD001 5mg/day + Glivec 600mg/day (Experimental): RAD001 5 mg was given in combination with Glivec/Gleevec 600mg/day.
  Interventions: Drug: RAD001; Drug: Imatinib 600mg/day (Glevec is the brand name for imatinib)
- Phase l: RAD001 2.5mg/day + Glivec 800mg/day (Experimental): RAD001 2.5 mg was given in combination with Glivec/Gleevec 800mg/day.
  Interventions: Drug: RAD001; Drug: Imatinib 600mg/day (Glevec is the brand name for imatinib)
- Phase ll - Stratum l (first-line resistant/refractory): RAD001 2.5mg/day + Glivec 600mg/day (Experimental): All first-line resistant/refractory patients received RAD001 2.5mg/day in combination with Glivec/Gleevec at a dose of 600mg/day.
  Interventions: Drug: RAD001; Drug: Imatinib 800mg/day (Glevec is the brand name for imatinib)
- Phase ll - Stratum ll: (post second-line therapy): RAD001 2.5mg/day + Glivec 600mg/day (Experimental): All post-second-line patients received RAD001 2.5mg/day in combination with Glivec/Gleevec at a dose of 600mg/day
  Interventions: Drug: RAD001; Drug: Imatinib 800mg/day (Glevec is the brand name for imatinib)

INTERVENTIONS:
Drug: RAD001 — RAD001 was in tablets of 0.5 mg, 1.0 mg, 2.5 mg and 5.0 mg strength and was taken by mouth, once a week or once a day depending upon the treatment group the patient was enrolled into.
  Other Names: everolimus
Drug: Imatinib 600mg/day (Glevec is the brand name for imatinib) — Glivec/Gleevec was supplied as commercialized 100 mg and 400 mg tablets. Gleevec/Glivec was provided as capsules of 100 mg strength in bottles containing 60 capsules each. The use of this supply was study center specific. Glivec/Gleevec was taken, by mouth, at a dose of 300 mg twice a day. The Glivec/Gleevec regimen was changed from 600 mg once a day to 300 mg BID, by an amendment since taking too many tablets at once was difficult for patients with gastro-intestinal disease. In the phase II part of the study all patients received Glivec 600 mg/day.
  Other Names: STI571
  Arms: Phase l: RAD001 2.5mg/day + Glivec 600mg/day; Phase l: RAD001 2.5mg/day + Glivec 800mg/day; Phase l: RAD001 5mg/day + Glivec 600mg/day
Drug: Imatinib 800mg/day (Glevec is the brand name for imatinib) — Glivec/Gleevec was supplied as commercialized 100 mg and 400 mg tablets. Gleevec/Glivec was provided as capsules of 100 mg strength in bottles containing 60 capsules each. The use of this supply was study center specific. Glivec/Gleevec was taken, by mouth. In the phase II part of the study all patients received Glivec 600 mg/day, except for 2 patients who received Glivec at a dose of 800 mg/day. This dose was permitted in Phase II as it was found to be safe in Phase I.
  Other Names: STI571
  Arms: Phase ll - Stratum l (first-line resistant/refractory): RAD001 2.5mg/day + Glivec 600mg/day; Phase ll - Stratum ll: (post second-line therapy): RAD001 2.5mg/day + Glivec 600mg/day

SUMMARY:
This trial was a Phase I/II, non-randomized, open label, multi-center study, following a sequential 2-part design.

DETAILED DESCRIPTION:
The first part, Phase I, was designed to assess whether there is a pharmacokinetic interaction between Glivec/Gleevec (imatinib) and RAD001(everolimus) as well as to collect safety data when these two drugs are co-administered. The second part, (Phase II), was designed to assess the potential efficacy of the combination in imatinib-resistant GIST patients in two strata of patients:

* Patients resistant to imatinib as first-line drug therapy and in whom the maximum tolerated dose was at least 600 mg/d (Stratum 1, first-line resistant/refractory)
* Patients resistant to imatinib as well as to post-imatinib drug therapy (Stratum 2, post second-line therapy).

It was decided to discontinue the study and close to further enrollment based on alternative treatment options that became available. Phase 1 and Phase 2 Stratum 1 were ended early on 02-Nov-2006. Investigators were allowed to complete the enrollment in the Phase 2 Stratum 2.

ELIGIBILITY:
Inclusion Criteria:

Phase l:

* Patients aged ≥ 18 years
* Patients with a histologically proven diagnosis of GIST and clinical evidence of resistance to imatinib despite at least 4 months continuous treatment with imatinib
* Patients with at least 2 months at a dosage of ≥ 600 mg/day (progression despite uninterrupted therapy for 2 months at ≥800 mg/d for patients entering the Phase I cohort investigating the 800 mg/d dose)
* Patients were to have at least one measurable lesion (longest diameter ≥20 mm on conventional CT or MRI scan
* patients were to have ≥10 mm on spiral CT) and were to have a WHO Performance Status Score ≤ 2.
* Patients also were to have adequate bone marrow, liver and renal function on imatinib treatment, as specified in the protocol

Phase ll:

• For Phase II (Stratum 2) patients must have progression on other 2nd line drug therapies following prior progression on imatinib (Stratum 2)

Exclusion Criteria:

* Women who are pregnant or breast-feeding
* Patients presenting with known or symptomatic CNS metastases or leptomeningeal involvement
* Patients with any concurrent major medical condition liable to compromise the patient's participation in the study (e.g. known HIV infection, uncontrolled diabetes, serious cardiac dysrhythmia or condition, New York Heart Association classification of III or IV, congestive cardiac failure, myocardial infarction with 6 months, unstable angina, chronic or acute renal or liver disease, uncontrolled infections including abscess or fistulae, etc.)
* Patients with a history of another malignancy within 5 years prior to study entry, except curatively treated non-melanotic skin cancer or in-situ cervical cancer
* Patients unwilling to or unable to comply with the protocol
* Patients who are receiving glucocorticoids (only if the p70s6 kinase1 assay is being performed), since these have been shown to inhibit p70s6 kinase1 activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2002-11-13 (Actual); Primary Completion 2008-09-03 (Actual); Study Completion 2008-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- United States (3):
  - Dana Farber Cancer Institute Dept of Sarcoma Oncology, Boston, Massachusetts
  - College of Physicians and Surgeons of Columbia University, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- Belgium (2):
  - Novartis Investigative Site, Edegem, Antwerpen
  - Novartis Investigative Site, Leuven
- France (5):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Villejuif
- Germany (6):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Tübingen

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the triasl in line with applicable laws and regulations.
  This trial data will be available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was a Phase I/II study, following a sequential 2-part design. The 1st part was designed to assess whether there was a pharmacokinetic interaction between Glivec/Gleevec and RAD001. The 2nd part was designed to assess the potential efficacy of the combination in Glivec/Gleevec-resistant GIST patients in 2 strata of patients.
Pre-assignment Details: An estimated maximum of 130 patients was planned to be enrolled into the study. In Phase I, there were 42 patients enrolled. In Phase II, there were 75 patients enrolled. 3 patients were excluded from all analyses due to a major protocol violation.
Groups:
- Phase ll: Stratum ll (Post Second-line Therapy): All post second-line therapy patients received RAD001 2.5mg/day in combination with Glivec/Gleevec at a dose of 600mg/day.
Period: Phase l by Treatment
Arm/Group | Phase l: RAD001 20mg/Week | Phase l: RAD001 2.5mg/Day + Glivec 600mg/Day | Phase l: RAD001 5mg/Day + Glivec 600mg/Day | Phase l: RAD001 2.5mg/Day + Glivec 800mg/Day | Phase ll - Stratum l (First-line Resistant/Refractory): RAD001 2.5mg/Day + Glivec 600mg/Day | Phase ll: Stratum ll (Post Second-line Therapy)
Started | 13 | 13 | 5 | 11 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 13 | 13 | 5 | 11 | 0 | 0
Not completed — Adverse Event | 1 | 4 | 2 | 3 | 0 | 0
Not completed — Abnormal laboratory value(s) | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Abnormal test procedure result(s) | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Disease progression | 12 | 8 | 2 | 5 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 1 | 0 | 0
Period: Phase ll by Stratum
Arm/Group | Phase l: RAD001 20mg/Week | Phase l: RAD001 2.5mg/Day + Glivec 600mg/Day | Phase l: RAD001 5mg/Day + Glivec 600mg/Day | Phase l: RAD001 2.5mg/Day + Glivec 800mg/Day | Phase ll - Stratum l (First-line Resistant/Refractory): RAD001 2.5mg/Day + Glivec 600mg/Day | Phase ll: Stratum ll (Post Second-line Therapy)
Started | 0 | 0 | 0 | 0 | 28 | 47
Completed | 0 | 0 | 0 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 28 | 46
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 10
Not completed — Abnormal laboratory values | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Disease progression | 0 | 0 | 0 | 0 | 23 | 31
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat population (ITT-population) consists of all patients who received at least one dose of RAD001 or Glivec/Gleevec in accordance to the study protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase l: RAD001 20mg/Week | Phase l: RAD001 2.5mg/Day + Glivec 600mg/Day | Phase l: RAD001 5mg/Day + Glivec 600mg/Day | Phase l: RAD001 2.5mg/Day + Glivec 800mg/Day | Phase ll - Stratum l (First-line Resistant/Refractory): RAD001 2.5mg/Day + Glivec 600mg/Day | Phase ll: Stratum ll (Post Second-line Therapy) | Total
Number analyzed (Participants) | 13 | 13 | 5 | 11 | 28 | 47 | 117
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The Intent-to-treat population (ITT-population) consists of all patients who received at least one dose of RAD001 or Glivec/Gleevec in accordance to the study protocol.
  Years
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 28 | 47 | 75
    (all) |  |  |  |  | 55.6 (13.16) | 59.3 (12.54) | 57.9 (12.81)
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The Intent-to-treat population (ITT-population) consists of all patients who received at least one dose of RAD001 or Glivec/Gleevec in accordance to the study protocol.
  Years
    number analyzed (Participants) | 13 | 13 | 5 | 11 | 0 | 0 | 42
    (all) | 53.5 (5.25) | 52.2 (14.11) | 53.8 (11.95) | 61.9 (13.25) |  |  | 55.3 (11.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 4 | 2 | 7 | 16 | 34
  Male | 11 | 10 | 1 | 9 | 21 | 31 | 83
Race/Ethnicity, Customized [Number; unit: Participants] — Population: The Intent-to-treat population (ITT-population) consists of all patients who received at least one dose of RAD001 or Glivec/Gleevec in accordance to the study protocol.
  Participants
    Caucasian | 13 | 12 | 5 | 11 | 27 | 47 | 115
    Black | 0 | 1 | 0 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs): Phase I & II
Description: Assessed safety and tolerability of the combination administration of RAD001 and imatinib when given to patients with imatinib-refractory gastro-intestinal stromal tumors (GIST) by number of participants with adverse events.
Time Frame: 4 - 8 weeks
Population: Safety Population: All patients (except for the 3 patients who did not meet the protocol inclusion/exclusion criteria) were included in the Safety population for Phase I. All patients were included in the Safety population for Phase II.
Measure: Number; unit: Participants
Arm/Group | Phase l: RAD001 20mg/Week | Phase l: RAD001 2.5mg/Day + Glivec 600mg/Day | Phase l: RAD001 5mg/Day + Glivec 600mg/Day | Phase l: RAD001 2.5mg/Day + Glivec 800mg/Day | Phase ll - Stratum l (First-line Resistant/Refractory): RAD001 2.5mg/Day + Glivec 600mg/Day | Phase ll: Stratum ll (Post Second-line Therapy)
Number analyzed (Participants) | 13 | 13 | 5 | 11 | 28 | 47
Participants | 13 | 13 | 5 | 11 | 27 | 47

2. Primary Outcome: Best Overall Response (BOR) as Assessed by Overall Response (Complete Response (CR) & Partial Response (PR)) - Phase I & II
Description: Assessed clinical efficacy of the combination regimen in this patient population per BOR by Overall response (CR + PR). Complete response: Disappearance of all target lesions; Partial response: ≥ 30% decrease in the sum of the longest diameter of target lesions compared to baseline (and not ≥20% increase compared to smallest sum).
Time Frame: 6 - 8 weeks
Population: Intent-to-treat (ITT) population: All patients (except for the 3 patients who did not meet the protocol inclusion/exclusion criteria) were included in the ITT population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase l: RAD001 20mg/Week | Phase l: RAD001 2.5mg/Day + Glivec 600mg/Day | Phase l: RAD001 5mg/Day + Glivec 600mg/Day | Phase l: RAD001 2.5mg/Day + Glivec 800mg/Day | Phase ll - Stratum l (First-line Resistant/Refractory): RAD001 2.5mg/Day + Glivec 600mg/Day | Phase ll: Stratum ll (Post Second-line Therapy)
Number analyzed (Participants) | 13 | 13 | 5 | 11 | 28 | 47
Percentage of Participants | 0 [0.0 to 0.0] | 1 [0.2 to 36.0] | 0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 1 [0.1 to 11.3]

3. Primary Outcome: Trough Concentrations for RAD001 and for Imatinib - Phase II
Description: Assessed the pharmacokinetics (PK) of the combination administration of RAD001 and imatinib in this patient population.
Time Frame: Part II Daily regimen: Baseline, Days 8, 15 and thereafter approximately every two months starting at month 3 whenever possible
Population: Pharmacokinetics (PK) population: The PK population included 18% of Stratum I patients and 47% of Stratum II patients
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Phase ll - Stratum l (First-line Resistant/Refractory): RAD001 2.5mg/Day + Glivec 600mg/Day | Phase ll: Stratum ll (Post Second-line Therapy)
Number analyzed (Participants) | 5 | 22
ng/mL
  Week 2: RAD001: number analyzed (Participants) | 1 | 5
  Week 2: RAD001 | 24.300 [24.30 to 24.30] | 12.100 [5.80 to 17.20]
  Week 3: RAD001: number analyzed (Participants) | 1 | 4
  Week 3: RAD001 | 19.900 [19.90 to 19.90] | 12.750 [7.62 to 23.30]
  Week 9: RAD001: number analyzed (Participants) | 0 | 2
  Week 9: RAD001 |  | 10.950 [10.40 to 11.50]
  Month 4: RAD001: number analyzed (Participants) | 0 | 3
  Month 4: RAD001 |  | 7.840 [6.90 to 10.30]
  Baseline: Imatinib: number analyzed (Participants) | 1 | 8
  Baseline: Imatinib | 472.00 [472.0 to 472.0] | 501.50 [402.0 to 1210.0]
  Week 2: Imatinib: number analyzed (Participants) | 2 | 15
  Week 2: Imatinib | 626.50 [549.0 to 704.0] | 540.00 [330.0 to 1970.0]
  Week 3: Imatinib: number analyzed (Participants) | 3 | 14
  Week 3: Imatinib | 572.00 [203.0 to 590.0] | 718.00 [412.0 to 4040.0]
  Week 9: Imatinib: number analyzed (Participants) | 0 | 6
  Week 9: Imatinib |  | 899.0 [295.0 to 1780.0]
  Month 4: Imatinib: number analyzed (Participants) | 1 | 7
  Month 4: Imatinib | 333.00 [333.0 to 333.0] | 446.00 [89.9 to 1350.0]
  Month 6: Imatinib: number analyzed (Participants) | 1 | 1
  Month 6: Imatinib | 181.00 [181.0 to 181.0] | 2040.00 [2040.0 to 2040.0]
  Month 8: Imatinib: number analyzed (Participants) | 0 | 2
  Month 8: Imatinib |  | 575.00 [566.0 to 584.0]
  Month 12: Imatinib: number analyzed (Participants) | 0 | 1
  Month 12: Imatinib |  | 324.00 [324.0 to 324.0]

4. Primary Outcome: Overall Survival (OS) - Phase I & II
Description: Assessed clinical efficacy of the combination regimen in this patient population per Overall Survival (OS). Overall survival was defined as the time from date of start of treatment to date of death due to any cause. For patients still receiving study medication at the time of the analysis, survival was censored at the date of last examination. If a patient was not known to have died but was no longer continuing with study medication, survival was censored at the date of last contact.
Time Frame: about 60 months
Population: ITT population: All patients (except for the 3 patients who did not meet the protocol inclusion/exclusion criteria) were included in the ITT population for phase I. All patients were included in the ITT population for phase II.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase l: RAD001 20mg/Week | Phase l: RAD001 5mg/Day + Glivec 600mg/Day | Phase l: RAD001 2.5mg/Day + Glivec 600mg/Day | Phase l: RAD001 2.5mg/Day + Glivec 800mg/Day | Phase ll - Stratum l (First-line Resistant/Refractory): RAD001 2.5mg/Day + Glivec 600mg/Day | Phase ll: Stratum ll (Post Second-line Therapy)
Number analyzed (Participants) | 13 | 13 | 5 | 11 | 28 | 47
months | 9.4 [5.6 to 13.8] | 10.9 [3.3 to NA] — NA - insufficient number of participants with events | 18.7 [3.8 to NA] — NA - insufficient number of participants with events | NA [12.0 to NA] — NA - insufficient number of participants with events | 14.9 [14.9 to NA] — NA - insufficient number of participants with events | 10.7 [6.3 to 16.8]

5. Secondary Outcome: mTOR Pathway Activity Before Treatment, and Inhibition of mTOR Pathway Activity During Treatment as a Predictive Factor of Response, as Shown by Molecular Pathological Examination of the Tumor.
Description: assess mTOR pathway activity before treatment, and inhibition of mTOR pathway activity during treatment as a predictive factor of response, as shown by molecular pathological examination of the tumor.
Time Frame: about 60 months
Population: Pharmacodynamic population: Molecular pathology and pharmacogenomic assessments were planned, but not carried out due to an alternative therapy that became available after the initiation of this study.
Arm/Group | Phase l: RAD001 20mg/Week | Phase l: RAD001 5mg/Day + Glivec 600mg/Day | Phase l: RAD001 2.5mg/Day + Glivec 600mg/Day | Phase l: RAD001 2.5mg/Day + Glivec 800mg/Day | Phase ll - Stratum l (First-line Resistant/Refractory): RAD001 2.5mg/Day + Glivec 600mg/Day | Phase ll: Stratum ll (Post Second-line Therapy)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Relationship Between Drug-induced Changes in the Principal Molecular Marker of Intratumoral mTOR Activity and Changes in Other Molecular Markers of Tumoral Activity (e.g. Indicators of Pathway Activity, Cell Proliferation and Apoptosis).
Description: assess the relationship between drug-induced changes in the principal molecular marker of intratumoral mTOR activity and changes in other molecular markers of tumoral activity (e.g. indicators of pathway activity, cell proliferation and apoptosis).
Time Frame: about 60 months
Population: as for outcome 5
Arm/Group | Phase l: RAD001 20mg/Week | Phase l: RAD001 5mg/Day + Glivec 600mg/Day | Phase l: RAD001 2.5mg/Day + Glivec 600mg/Day | Phase l: RAD001 2.5mg/Day + Glivec 800mg/Day | Phase ll - Stratum l (First-line Resistant/Refractory): RAD001 2.5mg/Day + Glivec 600mg/Day | Phase ll: Stratum ll (Post Second-line Therapy)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Relationship Between Drug-induced Changes in Tumoral Metabolism, as Shown by Functional Imaging With 18F-fluorodeoxyglucose Positron Emission Tomography (FDC-PET), With Clinical Outcome and Changes in Molecular Pathology.
Description: assess the relationship between drug-induced changes in tumoral metabolism, as shown by functional imaging with 18F-fluorodeoxyglucose positron emission tomography (FDC-PET), with clinical outcome and changes in molecular pathology.
Time Frame: about 60 months
Population: PET scans at baseline and as follow-up were planned to assess functional changes in tumors for patients on treatment. This analysis was not carried out due to alternative therapy that became available after the initiation of this study.
Arm/Group | Phase l: RAD001 20mg/Week | Phase l: RAD001 5mg/Day + Glivec 600mg/Day | Phase l: RAD001 2.5mg/Day + Glivec 600mg/Day | Phase l: RAD001 2.5mg/Day + Glivec 800mg/Day | Phase ll - Stratum l (First-line Resistant/Refractory): RAD001 2.5mg/Day + Glivec 600mg/Day | Phase ll: Stratum ll (Post Second-line Therapy)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: 4-Month Progression-free Survival (PFS) Rate - Phase II
Description: Assessed clinical efficacy of the combination regimen in this patient population per Progression-free survival (PFS). Progression-free survival (PFS) was the time from date of start of treatment to the date of first documented progression or death due to any cause. Per protocol (PP) population includes patients with no known overall lesion response during 4 months +/- 2 weeks, or who later had response of CR/PR/stable disease (SD). PP population excludes patients with no known response during 4 months + / -2 weeks and no subsequent CR/PR/SD.
Time Frame: about 4 months
Population: Per Protocol population: The per-protocol population included 82% of Stratum I patients and 75% of Stratum II patients.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase ll - Stratum l (First-line Resistant/Refractory): RAD001 2.5mg/Day + Glivec 600mg/Day | Phase ll: Stratum ll (Post Second-line Therapy)
Number analyzed (Participants) | 23 | 35
Percentage of participants | 17.4 [5.0 to 38.8] | 37.1 [21.5 to 55.1]

9. Primary Outcome: Progression-free Survival (PFS) - Phase II
Description: Assessed clinical efficacy of the combination regimen in this patient population per Progression-free survival (PFS). Progression-free survival (PFS) was the time from date of start of treatment to the date of first documented progression or death due to any cause. If a patient had not progressed or died, progression-free survival was censored at the time of last adequate tumor assessment.
  According to the study protocol no tumor assessments were performed after discontinuation of treatment with study drug. Therefore, for all patients who discontinued treatment without a documented progression but died thereafter, death was considered as PFS event only if it occurred within the regular safety follow-up of 28 days after discontinuation. Otherwise, the PFS time was censored at the last adequate tumor assessment.
Time Frame: about 60 months
Population: ITT population: All patients were included in the ITT population for Phase II.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase ll - Stratum l (First-line Resistant/Refractory): RAD001 2.5mg/Day + Glivec 600mg/Day | Phase ll: Stratum ll (Post Second-line Therapy)
Number analyzed (Participants) | 28 | 47
months | 1.9 [1.8 to 3.7] | 3.5 [1.9 to 5.2]

10. Post Hoc Outcome: All Collected Deaths
Description: On treatment deaths were collected from FPFT up to 28 days after study drug discontinuation, for a maximum duration of 35.52 months (treatment duration ranged from 0.36 to to 35.52 months for the phase I part) and a maximum duration of 21.88 months (treatment duration of 0.16 to 21.88 months for the phase II part). Deaths post treatment survival follow up were collected after the on treatment period, up to 70 months.
Time Frame: approx. 35.52 months, approx. 70 months
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Phase l: RAD001 20mg/Week | Phase l: RAD001 2.5mg/Day + Glivec 600mg/Day | Phase l: RAD001 5mg/Day + Glivec 600mg/Day | Phase l: RAD001 2.5mg/Day + Glivec 800mg/Day | Phase ll - Stratum l (First-line Resistant/Refractory): RAD001 2.5mg/Day + Glivec 600mg/Day | Phase ll: Stratum ll (Post Second-line Therapy)
Number analyzed (Participants) | 13 | 13 | 5 | 11 | 28 | 47
Participants
  Total Deaths | 12 | 8 | 3 | 3 | 9 | 22
  Deaths on-treatment | 2 | 3 | 0 | 2 | 3 | 6

ADVERSE EVENTS:
Time Frame: On-treatment deaths were collected from FPFT up to 28 days after study drug discontinuation, for a maximum duration of 35.52 months (treatment duration ranged from 0.36 to to 35.52 months for Phase I part) and a maximum duration of 21.88 months (treatment duration of 0.16 to 21.88 months for the Phase II part).
Description: Adverse Event: Any sign or symptom that occurs during the study treatment plus 28 days post treatment.
Groups:
- Phase I - RAD001 20mg/Week ++ Glivec 600mg/Day: RAD001 20 mg was given in combination with Glivec/Gleevec 600mg/day
- Phase I: RAD001 2.5mg/Day + Glivec 600mg/Day: RAD001 2.5 mg was given in combination with Glivec/Gleevec 600mg/day.
- Phase I: RAD001 5mg/Day + Glivec 600mg/Day: RAD001 5 mg was given in combination with Glivec/Gleevec 600mg/day.
- Phase I: RAD001 2.5mg/Day + Glivec 800mg/Day: RAD001 2.5 mg was given in combination with Glivec/Gleevec 800mg/day.
Arm/Group | Phase I - RAD001 20mg/Week ++ Glivec 600mg/Day | Phase I: RAD001 2.5mg/Day + Glivec 600mg/Day | Phase I: RAD001 5mg/Day + Glivec 600mg/Day | Phase I: RAD001 2.5mg/Day + Glivec 800mg/Day | Phase ll - Stratum l (First-line Resistant/Refractory): RAD001 2.5mg/Day + Glivec 600mg/Day | Phase ll: Stratum ll (Post Second-line Therapy)
Serious Adverse Events (participants affected / at risk) | 4/13 | 7/13 | 3/5 | 7/11 | 11/28 | 25/47
Other Adverse Events (participants affected / at risk) | 13/13 | 12/13 | 5/5 | 11/11 | 27/28 | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I - RAD001 20mg/Week ++ Glivec 600mg/Day (N=13) | Phase I: RAD001 2.5mg/Day + Glivec 600mg/Day (N=13) | Phase I: RAD001 5mg/Day + Glivec 600mg/Day (N=5) | Phase I: RAD001 2.5mg/Day + Glivec 800mg/Day (N=11) | Phase ll - Stratum l (First-line Resistant/Refractory): RAD001 2.5mg/Day + Glivec 600mg/Day (N=28) | Phase ll: Stratum ll (Post Second-line Therapy) (N=47)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 2 | 0 | 1 | 8
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 2
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 4
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 1 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Catheter related complication (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 3
Drug interaction (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 1 | 1 | 2 | 0 | 1 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mucosal haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 1 | 1
Ulcer haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Morganella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 4 | 2 | 0 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Costovertebral angle tenderness (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pelvic discomfort (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemodynamic instability (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I - RAD001 20mg/Week ++ Glivec 600mg/Day (N=13) | Phase I: RAD001 2.5mg/Day + Glivec 600mg/Day (N=13) | Phase I: RAD001 5mg/Day + Glivec 600mg/Day (N=5) | Phase I: RAD001 2.5mg/Day + Glivec 800mg/Day (N=11) | Phase ll - Stratum l (First-line Resistant/Refractory): RAD001 2.5mg/Day + Glivec 600mg/Day (N=28) | Phase ll: Stratum ll (Post Second-line Therapy) (N=47)
Anaemia (Blood and lymphatic system disorders) | 6 | 7 | 3 | 4 | 12 | 22
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 5 | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 5 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 2 | 2 | 4 | 7
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cyanosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 2 | 1 | 0 | 0 | 6
Eye oedema (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 1
Eye swelling (Eye disorders) | 1 | 0 | 0 | 0 | 2 | 1
Eyelid oedema (Eye disorders) | 0 | 2 | 0 | 4 | 4 | 8
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1
Orbital oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 5 | 2 | 3 | 11 | 12
Abdominal pain lower (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2 | 5
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 2
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 2 | 2 | 1 | 5 | 7
Diarrhoea (Gastrointestinal disorders) | 8 | 5 | 2 | 7 | 12 | 17
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 2 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2 | 0 | 3 | 6 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 1 | 3
Lip oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 7 | 8 | 5 | 7 | 12 | 16
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Painful defaecation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 2 | 1 | 3 | 4 | 7
Vomiting (Gastrointestinal disorders) | 3 | 3 | 3 | 5 | 6 | 14
Asthenia (General disorders) | 1 | 3 | 0 | 0 | 5 | 7
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 4
Chills (General disorders) | 0 | 0 | 0 | 2 | 1 | 2
Face oedema (General disorders) | 0 | 1 | 0 | 1 | 2 | 3
Fatigue (General disorders) | 9 | 8 | 2 | 9 | 15 | 16
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 1 | 3
General physical health deterioration (General disorders) | 1 | 0 | 2 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 2 | 2
Malaise (General disorders) | 1 | 0 | 0 | 0 | 1 | 1
Mucosal inflammation (General disorders) | 0 | 2 | 0 | 2 | 0 | 6
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0 | 4 | 5
Oedema peripheral (General disorders) | 2 | 2 | 1 | 8 | 8 | 17
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Pitting oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 5 | 3 | 3 | 4 | 9
Temperature intolerance (General disorders) | 0 | 2 | 0 | 0 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 4
Campylobacter infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis infective (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 2
Genital infection fungal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Helicobacter infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 4 | 3 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 3
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 2 | 2 | 1 | 3
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 4 | 0 | 1 | 0 | 4 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 1 | 2 | 2
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0
Weight decreased (Investigations) | 4 | 3 | 3 | 2 | 6 | 8
Weight increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 4 | 5 | 2 | 5 | 6 | 16
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 5 | 5 | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypovitaminosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Magnesium deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tetany (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 1 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mastication disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 0 | 4 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 1 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 4
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 2 | 1
Ageusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 2 | 0 | 1 | 4 | 2
Headache (Nervous system disorders) | 4 | 0 | 0 | 1 | 8 | 6
Hyposmia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 5
Distractibility (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 1 | 3 | 2 | 1 | 3
Nervousness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 1
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 2 | 3 | 1
Bladder spasm (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 2 | 1
Micturition frequency decreased (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 0 | 0
Nipple pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia of genital male (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pelvic discomfort (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Prostatic intraepithelial neoplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 1 | 2 | 3 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 2 | 1 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 2 | 5
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 2 | 6
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1 | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 3
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Periorbital oedema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2 | 2 | 4
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 1 | 1 | 2 | 5 | 13
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin fragility (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.